CLINICAL TRIAL: NCT01453673
Title: Results of Knee Arthroscopic Surgery for Treatment of Cruciate Ligament and Meniscus
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Tai-Yuan Chuang, doctor, Taipei Medical University WanFang Hospital
Other Study IDs: 100014
Record Dates: First submitted 2011-10-13; First posted 2011-10-18 (Estimated); Last update posted 2011-10-18 (Estimated); Status verified 2011-10

CONDITIONS: Knee Arthroscopic Surgery
Keywords: knee; Cruciate Ligament; Meniscus

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is a retrospective review of chart. Clinical results including range of motion, muscle power and scores will be recorded. Arthrocopic surgery of cruciate ligament and meniscus will be re-evaluated for clinical application.

ELIGIBILITY:
Inclusion Criteria:

* ACL reconstructions
* PCL reconstructions
* Meniscectomy or Meniscus repair

Exclusion Criteria:

* Open surgery for knee lesion
* Combined fracture or other associated injury around knee

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Knee Arthroscopic Surgery patients
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2011-05; Study Completion 2013-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Tai-Yuan Chuang, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan